CLINICAL TRIAL: NCT00844467
Title: Serotyping of Pneumococci
Brief Title: A Retrospective Epidemiological Study on Pneumococcal Infection in Children in Ministry of Health Hospital at EHSA Region in the Eastern Province
Acronym: IPD in saudi
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: King Saud University (Other)
Responsible Party: King saud university, King saud univ
Other Study IDs: king Saud university
Record Dates: First submitted 2009-02-10; First posted 2009-02-16 (Estimated); Last update posted 2009-02-16 (Estimated); Status verified 2009-02

CONDITIONS: Pneumococcal Infection
Keywords: Risk factors; Case fatality; disease burden; Resistance; Benefits of pneumococcal vaccination
MeSH Terms: conditions — Pneumococcal Infections | interventions — Serogroup

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

INTERVENTIONS:
Biological: serotypes and resistance — screening patients with invasive pneumococci

SUMMARY:
The purpose of this study is to establish retrospectively the incidence rates of invasive pneumococcal disease in children aged less than 5 years. The investigators allocate the El Hasa region for the study because it has higher incidence of sickle cell anemia. The study will include data from 2003 to 2007(before introduction of the vaccine) and then for 2008 and 2009 (after introduction of the vaccine).

DETAILED DESCRIPTION:
Data will be collected from patents files or records for 5 years before the introduction of the vaccine and for 2 years after the introduction of the vaccine. We assigned 4 doctors in each hospital to carry and supervise the work.

ELIGIBILITY:
Inclusion Criteria:

* Invasive pneumococcal disease
* Children under 5 years
* Children lived in Elhasa region

Exclusion Criteria:

* Children above 5 years
* No invasive pneumococcal disease

Ages: 3 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children under 5 years with invasive pneumococccal dis.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2009-02; Primary Completion 2009-10 (Estimated); Study Completion 2009-12 (Estimated)